CLINICAL TRIAL: NCT06946381
Title: CAMpania PugliA bRanch Iliaco
Acronym: CAMPARI
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Collaborators: University of Bari (Other)
Responsible Party: Principal Investigator, Umberto Marcello Bracale, Prof., Federico II University
Other Study IDs: CAMPARI
Record Dates: First submitted 2025-04-09; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Aortoiliac Aneurysm; Iliac Aneurysm
Keywords: evar; bevar; AAA
MeSH Terms: conditions — Iliac Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- MAIN: Consecutive patients treated with the e-liac device
  Interventions: Procedure: Evar

INTERVENTIONS:
Procedure: Evar — Branch Evar with the e-liac device

SUMMARY:
Spontaneus Multicentric Observational registry to investigate the medium and long-term performances of the Iliac E-liac Branch Device from Artivion for treatment of Aortoiliac aneurysms in a real-world consecutive patients cohort.

ELIGIBILITY:
Inclusion Criteria:

* An aortoiliac or aortic aneurysm of surgical interest based on the most recent local guidelines treated with the E-liac stent-graft system, alone or in combination with other devices

Exclusion Criteria:

* Patient's refusal to be enrolled in the registry
* Patient treated with devices not including the E-liac stent-graft system

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients feferred to the insitution
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Aneurysm related death | assessed after procedure at 30 days, 6 months, one year, two years, three years, four years, five years.
  Aneurysm related death
Procedure-related re intervention | assessed after procedure at 30 days, 6 months, one year, two years, three years, four years, five years
  Procedure-related re intervention

SECONDARY OUTCOMES:
Aneurysm sac dynamics | assessed after procedure at 30 days, 6 months, one year, two years, three years, four years, five years
  Variation in aneurysm sac diameter

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Azienda ospedaliero-universitaria consorziale policlinico di Bari, Bari, BA
  - Azienda Ospedaliera Universitaria Federico II, Naples

IPD SHARING:
Plan to Share IPD: No